CLINICAL TRIAL: NCT05527288
Title: Single-arm, Single-center, Non-randomized, Open-label Study on the Application of Amyloid Imaging Agent [18F]Florbetaben（18FBB） PET/CT Imaging to Distinguish Non-cognitively Impaired Subjects and Mild to Moderate Alzheimer Disease Subjects in Chinese Population
Brief Title: A Bridging Study on Efficacy and Safety of [18F]Florbetaben PET for Diagnosis of Alzheimer Disease Subjects in Chinese Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sinotau Pharmaceutical Group (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: YZGK-XT001
Record Dates: First submitted 2022-08-08; First posted 2022-09-02 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-09

CONDITIONS: Alzheimer Disease; Dementia; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Tauopathies; Neurodegenerative Diseases; Neurocognitive Disorders; Mental Disorders
Keywords: Florbetaben; Amyloid beta-protein; Alzheimer disease
MeSH Terms: conditions — Alzheimer Disease; Dementia; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Tauopathies; Neurodegenerative Diseases; Neurocognitive Disorders; Mental Disorders; Plaque, Amyloid | interventions — 4-(N-methylamino)-4'-(2-(2-(2-fluoroethoxy)ethoxy)ethoxy)stilbene

STUDY DESIGN:
Intervention Model Description: All eligible patients will receive a single administration of the imaging agent [18F]florbetaben at a radioactive dose of 300 MBq.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Non-cognitively impaired subjects or mild to moderate Alzheimer disease subjects (Experimental): Visually and quantitatively assess PET images obtained after single application of 300 MBq [18F]florbetaben and PET scanning of patients with healthy subjects and non-cognitively impaired subjects or mild to moderate Alzheimer disease subjects.
  Interventions: Drug: Drug: [18F]florbetaben

INTERVENTIONS:
Drug: Drug: [18F]florbetaben — All eligible patients will receive a single administration of the imaging agent [18F]florbetaben at a radioactive dose of 300 MBq.

SUMMARY:
This is a bridging study to visually and quantitatively assess PET images obtained after single application of 300 MBq [18F]florbetaben and PET scanning of patients with Alzheimer disease.

DETAILED DESCRIPTION:
This is a bridging study to visually and quantitatively assess PET images obtained after single application of 300 MBq [18F]florbetaben and PET scanning of patients with healthy subjects and non-cognitively impaired subjects or mild to moderate Alzheimer disease subjects. The diagnostic efficacy of the visual and quantitative assessments of 18FBB PET images for diagnosis of Alzheimer disease will be determined by comparison to the standard of truth (SoT) obtained through standard of care clinical diagnosis. Imaging results were compared with reference standards to assess the ability of 18FBB PET imaging to differentiate non-cognitively impaired subjects from mild to moderate AD subjects. To investigate the pharmacokinetic characteristics of healthy subjects after single intravenous administration of 18FBB in Chinese population. Verify the safety of subjects after a single intravenous administration of 18FBB in Chinese population.

ELIGIBILITY:
Inclusion Criteria:

1. Inclusion criteria for non-cognitively impaired subjects:

1. Male or female aged between 55 and 85 years old (including 55 and 85 years old);
2. The education level of primary school or above, and can cooperate with the tests required for research including neuropsychological tests (cognitive ability, language ability, visual and auditory acuity can meet the requirements of the test);
3. Be able to understand the purpose and experimental protocol of clinical research;
4. The researcher judges that the subjects are in good health, and there is no abnormal or abnormality in the comprehensive physical examination, vital sign examination and laboratory examination, but they can participate in this bridging clinical trial according to the judgment of the clinician;
5. Clinical dementia score (CDR) of 0, and the Mini-Mental State Examination Scale (MMSE score) of ≥28;
6. For women of potential fertility (not yet or within 2 years of menopause), effective contraceptive measures must be used during the study period and within 6 months after the end of the study (effective contraceptive measures refer to sterilization, intrauterine hormonal devices, contraception condoms, contraceptives/dose, abstinence or partner removal of the vas deferens, etc.); male subjects should agree to use contraceptives during the study period and within 6 months after the end of the study period;
7. Able to sign the informed consent form.

2. Inclusion criteria for subjects with mild to moderate AD:

1. Male or female aged between 55 and 85 years old (including 55 and 85 years old);
2. The education level of primary school or above, and the ability to complete the cognitive ability test and other tests stipulated in the program;
3. Diagnosed as probable AD according to NINCDS-ADRDA criteria;
4. 18≤MMSE score≤26;
5. CDR score of 0.5, 1 or 2;
6. The investigator judges that the subject's "caregiver" can provide accurate information and report on the patient's cognitive and functional abilities;
7. For women of potential fertility (not yet menopause or within 2 years of menopause), effective contraceptive measures must be used during the study period and within 6 months after the end of the study (effective contraceptive measures refer to sterilization, intrauterine hormonal devices, contraception condoms, contraceptives/dose, abstinence or partner removal of the vas deferens, etc.); male subjects should agree to use contraceptives during the study period and within 6 months after the end of the study period;
8. Able to sign the informed consent form.

3. Inclusion criteria for healthy subjects:

1. Male or female aged 18 to 40 years old (including 18 years old and 40 years old);
2. Good health or no major diseases, as judged by the investigator based on the following evaluations: medical history, vital signs, physical examination, electrocardiogram and results of clinical laboratory tests;
3. Not using any drugs;
4. EEG examination, judged as "normal";
5. Screening blood routine, blood biochemistry and urine routine are normal, or the abnormality has no clinical significance;
6. Women must use effective contraceptive measures during the study period and within 6 months after the end of the study (effective contraceptive measures refer to sterilization, intrauterine hormone devices, condoms, contraceptives/agents, abstinence or partner removal of the vas deferens, etc.) ; male subjects should agree to use contraception during the study period and within 6 months after the end of the study period;
7. Able to sign the informed consent form.

Exclusion Criteria:

1. Exclusion criteria for non-cognitively impaired subjects:

1. History of various mental illnesses such as anxiety disorders, affective disorders, and schizophrenia;
2. Depression Screening Scale (PHQ-9) of ≥ 5 points;
3. Anxiety Disorder Screening Scale (GAD-7) of ≥ 5 points;
4. Severe neurological diseases, such as cerebrovascular diseases, inflammatory or infectious diseases, or any metabolic encephalopathy, neurodegenerative diseases, including Parkinson's disease history or physical or imaging manifestations;
5. History of severe craniocerebral injury, craniocerebral surgery or intracranial hematoma with permanent brain injury;
6. The results of cranial magnetic resonance imaging (MRI) also meet the following imaging findings: ①There are two or more infarcts outside the brain stem (diameter greater than 2 cm); ②Key parts such as thalamus, hippocampus, entorhinal cortex and angular gyrus Lacunar infarction; ③Fazekas score of high white matter damage ≥3;
7. Brain MRI examination showed enlarged perivascular space with subcortical diameter >3mm in short axis;
8. SWI (susceptibility-weighted imaging) prompts: cerebral microbleeds ≥5 locations;
9. History of alcohol or drug abuse/dependence;
10. Contraindications of MRI examination: such as heart pacemaker or nerve stimulator or metal foreign body, high fever, etc.;
11. Invasive surgery is planned within one week after administration of the study drug;
12. Allergy to the investigational drug or any of its components and/or a history of severe allergic reaction to the drug or allergens (such as allergic asthma);
13. Any major disease or unstable disease state (such as unstable angina pectoris, myocardial infarction or coronary revascularization, heart failure, acute and chronic renal failure, chronic liver disease, severe lung disease, blood disease, poor blood sugar control, chronic infection in the past 2 years, received surgical treatment 7 days ago, advanced cardiac insufficiency (New York Heart Association (NYHA stage IV), etc.);
14. History of tumor within 5 years (except cervical carcinoma in situ, prostate carcinoma in situ or local skin cancer after surgery);
15. Human immunodeficiency virus (HIV), hepatitis C or Treponema pallidum antibody test positive, hepatitis B surface antigen positive (except hepatitis B carriers);
16. Received drug therapy or other treatments (such as chemotherapy) that cause large fluctuations in hematological or biochemical indicators or serious side effects within two weeks before the screening examination;
17. Receive any contrast agent or radiopharmaceutical within 48 hours before application of test drug, or will use contrast agent within 24 hours after administration of study drug;
18. Participated in clinical research of other drugs within 30 days before enrollment or within 5 half-lives of the study drug (whichever is longer), and/or used any radiopharmaceuticals before the administration of the study drug, and not more than 10 radioactive half-lives apart;
19. History of epilepsy;
20. History of electroconvulsive therapy;
21. Received medications that may affect cognition, such as anxiolytics, within 2 weeks prior to the screening exam, and a history of receiving antidepressants and/or antipsychotics;
22. History of delirium (e.g. after surgery);
23. Other investigators deem it inappropriate to participate in the trial.

2. Exclusion criteria for subjects with mild to moderate AD:

1. History of various serious mental illnesses (such as severe depression, anxiety, affective disorders, schizophrenia or schizoaffective disorder) with PHQ-9 ≥ 10 points or GAD-7 ≥ 10 points;
2. Epilepsy episode occurred within the past 1 year;
3. Dementia caused by other reasons or cognitive dysfunction caused by other reasons: such as vascular dementia, Parkinson's disease dementia, Lewy body dementia, normal intracranial pressure hydrocephalus, intracranial mass, central nervous system infection (Such as HIV, syphilis, etc.), metabolic encephalopathy, etc.;
4. The results of cranial MRI also meet the following imaging findings: ①There are more than two infarcts outside the brain stem (diameter greater than 2 cm); ②Lacunar infarction in key parts such as the thalamus, hippocampus, entorhinal cortex and angular gyrus ③The Fazekas score of high white matter damage ≥ 3;
5. Brain MRI examination showed enlarged perivascular space with subcortical diameter >3mm in short axis;
6. SWI prompt: cerebral microbleeds ≥5 locations;
7. History of alcohol or drug abuse/dependence;
8. Contraindications of MRI examination: such as heart pacemaker or nerve stimulator or metal foreign body, high fever, etc.;
9. Subjects who plan to undergo surgery and/or other invasive surgery within 24 hours after the application of the trial drug;
10. Allergy to the investigational drug or any of its components and/or history of severe allergic reaction to the drug or allergens (such as allergic asthma);
11. Any major disease or unstable disease state (such as unstable angina pectoris, myocardial infarction or coronary revascularization, heart failure, acute and chronic renal failure, chronic liver disease, severe lung disease, blood Diabetic patients with disease, poor blood sugar control, chronic infection in the past 2 years, received surgical treatment 7 days ago, advanced cardiac insufficiency (NYHA stage IV), major depressive episode, etc.);
12. History of tumor within 5 years (except cervical carcinoma in situ, prostate carcinoma in situ or local skin cancer after surgery);
13. HIV, hepatitis C or Treponema pallidum antibody test positive, hepatitis B surface antigen positive (except hepatitis B carriers);
14. History of physical examination or imaging examination of neurological diseases (such as severe cerebrovascular disease, inflammation, infectious diseases and degenerative diseases, etc.);
15. History of severe craniocerebral injury, craniocerebral surgery or intracranial hematoma with permanent brain injury;
16. Received drug therapy or other treatments (such as chemotherapy) that cause large fluctuations in hematological or biochemical indicators or serious side effects within two weeks before the screening examination;
17. Receive any contrast agent or radiopharmaceutical within 48 hours before application of test drug, or will use contrast agent within 24 hours after administration of test drug;
18. Participated in clinical research of other drugs within 30 days before enrollment or within 5 half-lives of the study drug (whichever is longer), and/or used any radiopharmaceuticals before the administration of the study drug, and not more than 10 radioactive half-lives apart;
19. Other investigators deem it inappropriate to participate in the trial.

3. Exclusion criteria for healthy subjects:

1. Any previous brain disease, such as cerebrovascular disease, inflammatory or infectious disease, or any neurodegenerative disease, including Parkinson's disease history or physical or imaging manifestations; history of traumatic brain injury or brain surgery or cranial Internal hematoma with a history of permanent brain injury;
2. Any previous major disease or unstable condition (such as unstable angina pectoris, dilated or hypertrophic cardiomyopathy, valvular heart disease, congenital heart disease, myocardial infarction or coronary revascularization, heart failure, chronic renal failure, Chronic liver disease, severe lung disease, blood disease, diabetes, chronic infection, epilepsy, history of mental illness);
3. Have used drugs in the past week;
4. HIV, hepatitis C or Treponema pallidum antibody test positive, hepatitis B surface antigen positive;
5. History of coagulation or coagulation disorder;
6. History of liver or gastrointestinal diseases or other conditions that interfere with drug absorption, distribution, excretion or metabolism determined by the investigator;
7. Past tumor history;
8. High risk of drug allergy (such as allergic asthma patients) or history of severe allergic reactions to allergens;
9. History of alcohol or drug abuse/dependence;
10. Significant occupational exposure to ionizing radiation (e.g. more than 50 mSv/year) or exposure to radioactive substances or ionizing radiation for therapeutic or research purposes within the past 10 years;
11. Received any drugs and treatments that may interfere with the test data or may cause serious side effects and are not completely washed out before enrollment, as judged by the investigator;
12. Pregnant or lactating women;
13. Hospitalization due to illness during the screening period;
14. Other investigators deem it inappropriate to participate in the trial.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-01-28 (Actual); Primary Completion 2021-09-12 (Actual); Study Completion 2021-09-12 (Actual)

PRIMARY OUTCOMES:
Verify the safety of subjects after a single intravenous administration of 18FBB in Chinese population. | Up to 4 weeks
  Safety will be evaluated by collection of Adverse Events.
Evaluation of the ability of qualitative readings of PET imaging to distinguish non-cognitively impaired subjects from mild to moderate AD subjects after a single intravenous administration of 18FBB in Chinese population. | Up to 4 weeks
  Sensitivity and specificity of18FBB PET images for diagnosis of Alzheimer disease will be measured by comparison to the standard of truth (SoT) obtained through standard of care clinical diagnosis.

SECONDARY OUTCOMES:
Evaluation of the ability of quantitative analysis of PET imaging to distinguish non-cognitively impaired subjects from mild to moderate AD subjects after a single intravenous administration of 18FBB in Chinese population. | Up to 4 weeks
  Sensitivity and specificity of 18FBB PET images for diagnosis of Alzheimer disease will be measured by comparison to the standard of truth (SoT) obtained through standard of care clinical diagnosis.
Measurement of the Maximum Plasma Concentration (Cmax) of healthy subjects after single intravenous administration of 18FBB in Chinese population. | Up to 4 weeks
  Pharmacokinetic characteristics is described by Cmax.
Measurement of the Peak Plasma Time (Tmax) of healthy subjects after single intravenous administration of 18FBB in Chinese population. | Up to 4 weeks
  Pharmacokinetic characteristics is described by Tmax.
Measurement of Area Under the Curve （AUC）for plasma concentration of healthy subjects after single intravenous administration of 18FBB in Chinese population. | Up to 4 weeks
  Pharmacokinetic characteristics is described by AUC.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No